CLINICAL TRIAL: NCT00180544
Title: A Prospective, Non-Randomized, Multicenter, Single-Arm, Clinical Trial to Assess the Safety and Efficacy of the RX HERCULINK 14 Peripheral Stent System for Treatment in de Novo or Restenotic Renal Artery Stenosis
Brief Title: Safety and Effectiveness Study of the HERCULINK 14 Stent to Treat Renal Artery Disease
Acronym: HERCULINK 14
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Device superceded by next generation device. Enrollment stopped, long term follow up was completed in August of 2004.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Maureen Kennedy, Abbott Vascular
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-707
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Renal Artery Obstruction
MeSH Terms: conditions — Renal Artery Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Male and female patients, who meet study eligibility criteria, agree to participate in the trial, and sign an informed consent, will be enrolled in the study. A HERCULINK™ 14 Peripheral Stent will be used in the treatment of suboptimal post- procedural percutaneous transluminal angioplasty (PTA) atherosclerotic renal artery stenoses.
  Interventions: Device: Stenting: Renal Artery

INTERVENTIONS:
Device: Stenting: Renal Artery — Male and female patients, who meet study eligibility criteria, agree to participate in the trial, and sign an informed consent, will be enrolled in the study. A HERCULINK™ 14 Peripheral Stent will be used in the treatment of suboptimal post- procedural percutaneous transluminal angioplasty (PTA) atherosclerotic renal artery stenoses.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the RX HERCULINK 14 Peripheral Stent System in treating atherosclerotic renal artery stenosis.

DETAILED DESCRIPTION:
A prospective, non-randomized, multi-center, single-arm clinical trial to evaluate the safety and efficacy of the RX HERCULINK™ 14 Peripheral Stent System in the treatment of suboptimal post- procedural percutaneous transluminal angioplasty (PTA) results in de novo or restenotic atherosclerotic renal artery stenoses.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of renal artery atherosclerosis; candidate for renal artery angioplasty and stenting; blood pressure >160/90

Exclusion Criteria:

* Totally occluded renal artery on the opposite side; only one functioning kidney; target lesion is in a transplanted kidney; renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2000-07; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Primary patency . | at 9-months

SECONDARY OUTCOMES:
Acute procedural success | Acute
Access site events requiring surgical repair or intervention | Acute
Major adverse events (e.g. death, nephrectomy, target lesion revascularization (TLR) | at 30 days
TLR | at 9 months
Renal function | measured at 1, 6, 9, and 12-month follow-up, and every three months thereafter until approximately May 2003 or until patient 169 completes 12 month follow-up.
Changes in blood pressure | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ramee, M.D., Principal Investigator — Alton Ochsner Medical Foundation
Locations (1):
- Alton Ochsner Medical Foundation, New Orleans, Louisiana, United States